CLINICAL TRIAL: NCT00488696
Title: Branched Stent-Graft Repair for Endo Repair of Aneurysms Involving the Proximal Aortic Arch
Brief Title: Branched Aortic Arch Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study team was unable to identify eligible subjects. The study is being closed out due to a lack of subject eligibility. Zero subjects were enrolled in the entire duration of the study.
Sponsor: Timothy Chuter, MD (Other)
Responsible Party: Sponsor-Investigator, Timothy Chuter, MD, Sub-Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-03930
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Aortic Aneurysm of the Proximal Arch
Keywords: Aneurysm; Aortic Arch; Endovascular; Stent-Graft
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional (Experimental): Endovascular Bifurcated Stent Graft: The investigational operation involves placing a stent-graft over the aortic aneurysm.
  Interventions: Device: Endovascular Bifurcated Stent-Graft

INTERVENTIONS:
Device: Endovascular Bifurcated Stent-Graft — Treatment of Aneurysm involving the proximal aortic arch with endovascular bifurcated stent-graft.

SUMMARY:
This is a study to assess the safety and effectiveness of endovascular treatment of aortic aneurysms involving the proximal aortic arch. The investigational operation involves placing a stent-graft over the aortic aneurysm.

DETAILED DESCRIPTION:
An aneurysm is a localized bulge in the wall of an artery. Aneurysms of the aorta are prone to progressive dilatation, which if left untreated ultimately results in rupture, internal bleeding and death. Traditional open surgery involves aortic exposure through a long incision, aortic clamping to interrupt blood flow, and replacement or repair of the dilated aortic segment using a fabric conduit (graft), which is sutured (anastomosis) to the nondilated arteries above and below the aneurysm. Some subjects are able to withstand such a large operation better than others, but many suffer complications, and all suffer pain, debility, and a lengthy stay in hospital.

Endovascular aneurysm repair is a less invasive alternative that substitutes a trans-arterial route to the aneurysm for direct exposure, and stent-mediated attachment for sutured anastomosis. Compared to open surgical repair, endovascular repair is associated with less physiological derangement, less pain, less blood loss, lower complication rates and shorter hospital stay. Consequently, endovascular repair has become standard therapy for aneurysms of the abdominal aorta and descending thoracic aorta, where there are no vital branches and endovascular exclusion rarely causes ischemic complications.

Open surgical repair of the proximal aortic arch requires hypothermic circulatory arrest, because it deprives the heart of its outflow and the brain of its inflow. Endovascular repair also obstructs outflow from the heart, but only for a few seconds, while the graft is released from its delivery sheath. The greater problem is inflow to the brain. In anticipation of aortic arch exclusion, the brachiocephalic circulation requires an alternative source of blood. One alternative is bypass from the ascending aorta. However, this requires median sternotomy and partial aortic clamping, both of with are potential sources of morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Aneurysm of the aortic arch larger than 6cm in diameter, or symptomatic aneurysm of the aortic arch, of any diameter, or any arch aneurysm with a 2-year rupture rate estimated to be more than 20%.
* Anticipated mortality rate with open repair estimated to be more than 20%.
* Suitable arterial anatomy for stent-graft
* Life expectancy more than 2 years
* Ability to give informed consent and willingness to comply with follow-up schedule

Exclusion Criteria:

* Free rupture of the aneurysm
* Pregnancy
* Anaphylactic reaction to contrast material
* Allergy to stainless steel or polyester
* Unwillingness or inability to comply with the follow-up schedule
* Serious systemic or groin infection
* Uncorrectable coagulopathy
* Significant presence of carotid artery atherosclerosis
* Arrhythmia define as 2nd- and 3rd-degree atrioventricular block or sinus node disease, such as sick sinus syndrome and symptomatic bradycardia, unless the patient already has a pacemaker in place and cardiology consultation confirms that it is safe to proceed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Actual)

PRIMARY OUTCOMES:
Successful implantation of bifurcated stent-graft for repair of Aneurysm involving the proximal aortic arch | 1 month

SECONDARY OUTCOMES:
Stability of bifurcated stent-graft for repair of Aneurysm involving the proximal aortic arch | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Linda M Reilly, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Division of Vascular and Endovascular Surgery, San Francisco, California, United States

REFERENCES:
- [Background] Svensson LG, Crawford ES, Hess KR, Coselli JS, Raskin S, Shenaq SA, Safi HJ. Deep hypothermia with circulatory arrest. Determinants of stroke and early mortality in 656 patients. J Thorac Cardiovasc Surg. 1993 Jul;106(1):19-28; discussion 28-31. PMID 8321002
- [Background] Ergin MA, Griepp EB, Lansman SL, Galla JD, Levy M, Griepp RB. Hypothermic circulatory arrest and other methods of cerebral protection during operations on the thoracic aorta. J Card Surg. 1994 Sep;9(5):525-37. doi: 10.1111/j.1540-8191.1994.tb00886.x. PMID 7994095
- [Background] Criado FJ, Barnatan MF, Rizk Y, Clark NS, Wang CF. Technical strategies to expand stent-graft applicability in the aortic arch and proximal descending thoracic aorta. J Endovasc Ther. 2002 Jun;9 Suppl 2:II32-8. PMID 12166839
- [Background] Saccani S, Nicolini F, Beghi C, Marcato C, Uccelli M, Larini P, Budillon AM, Agostinelli A, Gherli T. Thoracic aortic stents: a combined solution for complex cases. Eur J Vasc Endovasc Surg. 2002 Nov;24(5):423-7. doi: 10.1053/ejvs.2002.1687. PMID 12435342
- [Background] Chuter TA, Buck DG, Schneider DB, Reilly LM, Messina LM. Development of a branched stent-graft for endovascular repair of aortic arch aneurysms. J Endovasc Ther. 2003 Oct;10(5):940-5. doi: 10.1177/152660280301000517. PMID 14656176
- [Background] Schneider DB, Curry TK, Reilly LM, Kang JW, Messina LM, Chuter TA. Branched endovascular repair of aortic arch aneurysm with a modular stent-graft system. J Vasc Surg. 2003 Oct;38(4):855. doi: 10.1016/s0741-5214(03)01024-3. No abstract available. PMID 14560244